CLINICAL TRIAL: NCT05038124
Title: A Pilot Study to Assess the Safety and Efficacy of Preoperative Stereotactic Body Radiotherapy for the Treatment of Metastatic Disease in Bone Requiring Surgical Stabilization
Brief Title: A Study of Stereotactic Body Radiotherapy (SBRT) and Surgical Stabilization for People With Cancer That Has Spread to the Bone
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-216
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Cancer
Keywords: Skeletal metastases; Stereotactic Body Radiotherapy (SBRT); Surgical Stabilization; Bone cancer; 21-216
MeSH Terms: conditions — Neoplasm Metastasis; Bone Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a pilot study to evaluate the safety of preoperative stereotactic body radiotherapy (SBRT) with short-interval surgical stabilization.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative Stereotactic Body Radiotherapy (SBRT) (Experimental): Target lesions will be treated with preoperative SBRT consisting of biologically effective dose (BED10) of 50.4 - 81.6 Gy delivered in either three fractions or a single fraction. Active sparing of the intended surgical approach will be incorporated into the radiation plan by creating an avoidance structure. Surgical stabilization will proceed within 1 week of completion of radiotherapy. Pathologic specimens will be obtained intraoperatively via existing surgical access for histologic and molecular analysis. An optional research MRI with perfusion will be performed within 30 days prior to radiation simulation and within one-week after radiation therapy using 3T scanner. If patients receive radiation simulation at a non-MSK Manhattan site, MRI with Perfusion will not be performed.
  Interventions: Radiation: Preoperative Stereotactic Body Radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Preoperative Stereotactic Body Radiotherapy (SBRT) — Target lesions will be treated with preoperative SBRT consisting of biologically effective dose (BED10) of 50.4 - 81.6 Gy delivered in either three fractions or a single fraction.

SUMMARY:
The purpose of this study is to test the safety of stereotactic body radiation therapy (SBRT) followed by surgical stabilization within 1 week. All participants will have metastatic cancer in the bone (bone metastases), and they will be at risk of pathologic fracture (broken bone caused by a disease). Another purpose of this study is to see if the treatment approach of SBRT followed by surgical stabilization within 1 week prevents cancer from returning to the bone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic cancer with radiologic evidence of skeletal metastases
* Treatment target involving humerus, radius, pelvis, sacrum, femur, or tibial diaphysis
* Age at enrollment ≥18 years
* Life expectancy >3 months
* Ability to tolerate radiation simulation and treatment with immobilization of involved anatomic site
* Surgical candidate, as determined by the treatment team
* Ability to obtain informed consent from patient or legally authorized representative in the setting of patient with impaired decision-making capacity.
* Must agree to practice an effective contraceptive method (for those with reproductive potential)

Exclusion Criteria:

* Prior radiotherapy to the treatment site
* Prior surgery involving the treatment site
* Tumor volume or distribution precluding effective SBRT
* Expected skin dose at the operative site ≥9 Gy
* Imminently impending fracture requiring immediate stabilization surgery
* Involvement of proximal tibia
* Autoimmune connective tissue disorder
* Administration of radiosensitizing medication 3 days before, during, and 3 days after RT
* Active infection
* Absolute neutrophil count <1.0
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
risk of major wound complications | 6 weeks after preoperative SBRT
  Major wound complications are defined as reoperation for wound revision, clinically diagnosed surgical site infection, readmission for wound care, or prolonged (>3 weeks postoperatively) active wound care.

SECONDARY OUTCOMES:
rate of local control | 1 year
  Failure of local control is defined as a new lesion within the radiation or surgical field, significant progression of an existing lesion, or reoperation or reirradiation due to tumor progression.

CONTACTS AND LOCATIONS:
Overall Officials: Maksim Vaynrub, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All protocol activities), New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm